CLINICAL TRIAL: NCT01022463
Title: Effect of Ivabradine vs Atenolol on Heart Rate and Effort Tolerance in Patients With Mild to Moderate Mitral Stenosis and Normal Sinus Rhythm
Brief Title: Effect of Ivabradine on Heart Rate & Effort Tolerance in Mitral Stenosis in Sinus Rhythm
Acronym: IVA-MS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Dr Neeraj Parakh, Govind Ballabh Pant hospital, New Delhi, India
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F-2/IEC/MAMC/09/No.192
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2010-11

CONDITIONS: Mitral Stenosis
MeSH Terms: conditions — Mitral Valve Stenosis | interventions — Ivabradine; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine (Active Comparator): Crossover study to compare ivabradine and atenolol
  Interventions: Drug: Ivabradine; Drug: Atenolol
- Atenolol (Placebo Comparator)
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 5 mg BId for 4 weeks
  Arms: Ivabradine
Drug: Atenolol — 50 mg od for 4 weeks

SUMMARY:
The purpose of this study is to study the effect of Ivabradine vs Atenolol on heart rate and effort tolerance in patients with mild to moderate mitral stenosis and normal sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate mitral stenosis (Mitral valve area: 1.0 cm2 - 2.0 cm2 on echocardiography) with normal sinus rhythm
2. Age >18 years
3. Need for rate control therapy for symptoms

Exclusion Criteria:

1. Atrial fibrillation
2. Other significant valvular lesions (More than mild AS/AR/MR)
3. Denial of consent
4. Unable to do TMT/Contraindication for TMT
5. Need for surgical treatment or BMV
6. Presence of significant non-cardiac co-morbidities
7. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in effort tolerance ( in minutes/Mets) from baseline with the study drugs at the end of stipulated 4 weeks | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Neeraj Parakh, MD, DM, Principal Investigator — G. B. Pant Hospital, New Delhi
Locations (1):
- G. B. Pant Hospital, New Delhi, National Capital Territory of Delhi, India